CLINICAL TRIAL: NCT07369804
Title: Safety and Efficacy of Focused LED-Based Repeated Low-Level Red-Light Therapy in Myopic Adults: A Single-Arm Pilot Study
Brief Title: Study on Safety and Efficacy of Focused LED-Based Red-Light Therapy in Myopic Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20250606001
Record Dates: First submitted 2025-09-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Myopia; Red-Light Therapy; Light-Emitting Diode
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fLED-based red-light therapy (Experimental)
  Interventions: Device: fLED-based red-light therapy

INTERVENTIONS:
Device: fLED-based red-light therapy — Eligible subjects will receive fLED-based red-light therapy (650nm, 1500 lux, 0.20mW) administered twice daily (3-minute sessions per treatment, minimum 4-hour interval between sessions) over 5 consecutive weekdays, combined with SVS for a total of 28 days.

SUMMARY:
This research project is a prospective, single-arm, open-label pilot study designed to evaluate the efficacy and safety of focused LED-based repeated low-level red-light (fLED-RLRL) therapy in myopic adults. The primary objective is to assess whether the therapy can increase choroidal thickness and improve choroidal blood flow. The secondary objective is to evaluate the safety and tolerability of red light therapy in adult myopes.

The study will enroll 14 myopic adults aged 18 to 50 years, with spherical equivalent refractions ranging from -0.50 to -6.00 diopters. Participants will receive home-based fLED-RLRL therapy (wavelength 650 ± 10 nm, power 0.20 mW) twice daily for 3 minutes per session, 5 days per week, over a total of 28 days, combined with single-vision spectacles. The fLED red-light device employs a standard LED semiconductor chip integrated with a total internal reflection (TIR) lens and microlenses to deliver a precise and concentrated beam, enabling accurate focusing of light energy on the target area. A video tutorial will be provided to guide device usage, and support from the research team will be available throughout the study.

Before the treatment, baseline data will be collected from each participant. Baseline and follow-up assessments (days 7, 14, 21, 28) will include comprehensive ophthalmic examinations: visual acuity, intraocular pressure, slit-lamp examination, autorefraction and subjective refraction, optical coherence tomography (OCT), optical coherence tomography angiography (OCTA), and posterior blood flowgraphy. These assessments will monitor structural and functional changes in the retina and choroid, as well as adverse events (e.g., retinal damage, prolonged after-images).

Primary and secondary outcomes will include changes in choroidal thickness, choroidal blood flow, ocular biometric parameters, spherical equivalent refraction, and visual acuity. Additional imaging assessments, such as posterior blood flowgraphy, OCT, and OCTA scans, will also be evaluated.

This pilot study aims to preliminarily explore the safety and efficacy of an fLED red-light therapy system integrated with machine vision for myopia management by analyzing choroidal parameters over a short-term treatment period. By providing a safer alternative to current laser-based therapies, this project seeks to advance the field of myopia treatment, offering a novel solution that aligns with the increasing demand for effective and safe interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years.
2. SE refractions between -0.50 and -6.00 diopters (D)
3. Astigmatism of 1.50 D or less.
4. Best corrected monocular visual acuity better than 20/20 (Snellen equivalent).
5. Willingness to provide written informed consent and comply with the treatment protocol.

Exclusion Criteria:

1. Strabismus or binocular vision abnormalities in either eye.
2. Ocular abnormalities in either eye or other systemic abnormalities.
3. Previous or current use of myopia control interventions (e.g., orthokeratology, low-dose atropine, pirenzepine) within the past 6 months.
4. History of ocular surgeries (e.g., cataract surgery and LASIK/SMILE).
5. Afterimage time > 5 minutes (contraindications to RLRL therapy).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in choroidal thickness measured by OCT | Choroidal thickness will be measured on baseline, days 7, 14, 21, and 28 following treatment initiation.
  Optical coherence tomography (OCT) imaging will be performed using the ultra-wide field swept-source OCT system (VG200, SVision Imaging, Ltd., Luoyang, China) to measure subfoveal choroidal thickness (SFCT).

SECONDARY OUTCOMES:
Change in axial length (AL) measured by IOLMaster 700 | Axial length will be measured on baseline, days 7, 14, 21, and 28 following treatment initiation.
  Change in axial length (AL) will be measured by IOLMaster 700 (Carl Zeiss Meditec, Oberkochen, Germany) .
Change in Best corrected visual acuity (BCVA) using ETDRS chart | BCVA will be measured on baseline, days 7, 14, 21, and 28 following treatment initiation.
  An Early Treatment Diabetic Retinopathy Study (ETDRS) chart (Precision Vision, Villa Park, Illinois, USA) with standard illumination will be used to measure distance visual acuity. Best corrected visual acuity (BCVA) will be measured at 4 meters.
Change in SE measured by auto-refractor and subjective refraction | SE will be measured on days 28 following treatment initiation.
  Auto-refraction will be conducted using an auto-refractor (KR-8800, Topcon, Tokyo, Japan). The same auto-refractor will be used throughout the study. It will be calibrated before each examination session to ensure there is no equipment drift during the long follow-up process. Subjective refraction will be conducted by a trained optometrist using a phoropter or trial frame and lenses. The same equipment will be used throughout the study. It will be calibrated before each examination session to ensure reliability and accuracy of the refraction results during the long follow-up process.
Change in ocular posterior segment blood flow metrics on the LSFG-NAVI | Ocular posterior segment blood flow metrics will be measured on baseline, days 7, 14, 21, and 28 following treatment initiation.
  The Laser Speckle Flowgraphy system (LSFG-NAVI) will be utilized to assess blood flow metrics in the posterior segment of the eye. This method involves capturing and analyzing dynamic changes in speckle patterns created by laser light reflecting off moving blood cells, specifically targeting the retinal and choroidal blood flow.
Change in choroidal vascularity index (CVI) measured by OCTA | Change in choroidal vascularity index will be measured on baseline, days 7, 14, 21, and 28 following treatment initiation.
  Change in choroidal vascularity index (CVI) will be assessed by optical coherence tomography angiography (OCTA). OCTA imaging will be performed using the ultra-wide field swept-source OCTA system (VG200, SVision Imaging, Ltd., Luoyang, China). Two imaging sessions will be performed, including a peripapillary scan centered on the optic disc (ONH Angio6*6 512*512 R4 mode) and a perifoveal scan centered on the macula (Angio6*6 512*512 R4 mode), to detect any structural changes in the macula and optic nerve head.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No